CLINICAL TRIAL: NCT00237705
Title: Intravenous Metoclopramide for the Treatment of Post Concussive Headache: a Randomized Placebo Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vancouver General Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CO4-0025
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2006-12-05 (Estimated); Status verified 2006-12

CONDITIONS: Post Concussive Headache; Post Concussive Syndrome
Keywords: Headache; Concussion; Post concussive syndrome; Head trauma
MeSH Terms: conditions — Post-Concussion Syndrome; Headache; Brain Concussion; Craniocerebral Trauma | interventions — Metoclopramide

INTERVENTIONS:
Drug: metoclopramide

SUMMARY:
Concussion is defined as any temporary disturbance in brain function following a blow to the head. It may not involve a loss of consciousness and usually results in a post concussive headache (PCH) immediately after the injury. Between 30 and 50 percent of patients with concussion will develop postconcussive syndrome (PCS) consisting of symptoms such as headache, and a variety of other debilitating symptoms lasting several weeks to months.

The objective of this study is to determine if metoclopramide, a drug commonly used in the treatment of migraine headache, will be effective in relieving PCH and in preventing PCS.

Eligible patients will have a history of a concussion resulting in headache within the past 24 hours. Patients will rate their pain on a standard scale before and after being treated with one or two intravenous doses of either metoclopramide or saltwater placebo. They will be contacted by telephone 1, 4 and 8 weeks later in order to determine if they have developed the postconcussive syndrome.

DETAILED DESCRIPTION:
PURPOSE AND OBJECTIVES The primary objective of this study is to prospectively evaluate the effect of metoclopramide in ED patients with minor head injury. The primary hypothesis is that the administration of intravenous metoclopramide will be effective in relieving the symptoms of acute post traumatic headache in ED patients with minor head injury.

The secondary hypothesis is that the administration of intravenous metoclopramide will also be effective in reducing the incidence of chronic post-concussive syndrome in ED patients with minor head injury. The research question is "Does the administration of intravenous metoclopramide at a dose of 10 or 20 mg to adult ED patients experiencing headache following a minor head injury result in a significant decrease in pain severity as measured on a 10cm visual analogue scale, as compared to placebo?"

RESEARCH METHODOLOGY This is a prospective, double-blind, randomized, placebo-controlled trial.

Only patients who meet the following inclusion criteria will be recruited:

1. History of blunt head trauma within preceding 24 hours
2. Immediate and transient post traumatic impairment of neurological functions such as alteration of consciousness, amnesia, disorientation, or disturbance of vision or equilibrium.
3. Onset of headache within one hour of trauma.
4. Significant intra-cranial injury excluded by CT scan or clinical assessment.

Exclusion criteria will include age less than or equal to 16 years, known or suspected pregnancy, known hypersensitivity or intolerance to metoclopramide, inability to give informed consent, known gastrointestinal hemorrhage, perforation or obstruction, known seizure disorder, known pheochromocytoma, concurrent significant CNS depression due to drugs or alcohol, or concurrent treatment for psychiatric illness.

Patients will be randomized and asked to grade their headache pain severity on a 10-cm non-hatched visual analog scale (VAS) before the administration of the study drugs. They will then receive either 10 mg (2ml) of metoclopramide or 2 ml of saline placebo. After 15 minutes they will again complete the VAS. If their headache is not satisfactorily relieved they will be offered a second dose of study drug and the VAS will be completed again 30 minutes later. Patients will be contacted 1, 4 and 8 weeks later in order to complete a telephone questionnaire to assess for PCS symptoms.

The primary comparison will be between the proportion of patients achieving significant pain relief in each of the two study arms and a difference of 20% of greater in these proportions will be considered clinically significant. A t-test of two proportions will be used and p less than or equal to 0.05 will be considered statistically significant. Secondary outcomes will be evaluated for hypothesis generating purposes using appropriate parametric and non-parametric statistics with corrections for multiple comparisons as needed.

ELIGIBILITY:
Inclusion Criteria:

* Only patients who meet the following inclusion criteria will be recruited:

  1. History of blunt head trauma within preceding 24 hours.
  2. Immediate and transient post traumatic impairment of neurological functions defined as alteration of consciousness, amnesia, disorientation, disturbance of vision or equilibrium (10).
  3. Onset of headache within one hour of trauma.

Exclusion Criteria:

* Patients with any of the following exclusion criteria will not be enrolled:

  1. Age less than or equal to 19 years.
  2. Known or suspected pregnancy.
  3. Known hypersensitivity or intolerance to metoclopramide.
  4. Inability to give informed consent.
  5. Known gastrointestinal hemorrhage, perforation or obstruction.
  6. Known seizure disorder.
  7. Known pheochromocytoma.
  8. Concurrent significant CNS depression due to drugs or alcohol.
  9. Concurrent treatment for psychiatric illness.
  10. Any acute brain injury on CT scan (if performed) as defined by any radiographic finding which would normally require admission to hospital and neurological follow up

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-05

PRIMARY OUTCOMES:
The primary outcome of acute PCH relief will be determined by measuring the difference between VAS score at baseline and after the last dose of study drug.

SECONDARY OUTCOMES:
The secondary outcome of PCS will be measured by telephone questionnaire using the Rivermead Post Concussion Symptoms Questionnaire at 1, 4 and 8 weeks after injury

CONTACTS AND LOCATIONS:
Overall Officials: David W Harrison, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada